CLINICAL TRIAL: NCT06234423
Title: A Phase 1, First-in-Human Study of CUSP06, a Cadherin-6 (CDH6)-Directed Antibody-Drug Conjugate, in Patients With Platinum-Refractory/Resistant Ovarian Cancer and Other Advanced Solid Tumors
Brief Title: A Study of CUSP06 in Patients With Platinum-Refractory/Resistant Ovarian Cancer and Other Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: OnCusp Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CUSP06-1001
Record Dates: First submitted 2024-01-10; First posted 2024-01-31 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Cancer; Solid Tumor
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Exploratory Cohort 1 (Experimental)
  Interventions: Drug: CUSP06
- Expansion Cohort 1 (Experimental)
  Interventions: Drug: CUSP06
- Expansion Cohort 2 (Experimental)
  Interventions: Drug: CUSP06

INTERVENTIONS:
Drug: CUSP06 — Antibody drug conjugate (ADC)

SUMMARY:
This phase 1 study will evaluate the safety, tolerability, pharmacokinetics, and efficacy of CUSP06 in patients with platinum-refractory/resistant ovarian cancer and other advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided prior to any screening procedures.
* Male or female patients, ≥18 years of age at the time of obtaining informed consent.
* Patients with histologically or cytologically confirmed advanced solid tumors previously treated with standard of care systemic therapy, or for whom no standard therapy is available.
* Willingness to provide archival tumor tissue, when available. If no archival tissue is available, willingness to undergo a pretreatment biopsy if medically feasible and safe.
* Measurable disease per RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 and life expectancy of ≥12 weeks.
* Adequate organ function as defined by:

  * Absolute neutrophil count (ANC) ≥1.5 x 109/L (1500/µL), without colony-stimulating factor support for the past 14 days.
  * Platelets ≥100.0 x 109/L (100 000/µL).
  * Hemoglobin ≥9.0 g/dL (without blood transfusion in 2-week period prior to screening).
  * Creatinine clearance (CrCl) ≥45 mL/min as calculated by the Cockcroft-Gault method.
  * Serum total bilirubin ≤ 1.5 x the upper limit of normal (ULN).
  * Aspartate aminotransferase (AST) ≤2.5 x ULN; alanine aminotransferase (ALT) ≤ 2.5 x ULN.
  * International normalized ratio (INR) ≤ 1.5; activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN.
  * Left ventricular ejection fraction (LVEF) ≥50% as per echocardiography (ECHO) or multi-gated acquisition scan (MUGA).
  * Q wave to T wave (QT) interval corrected for heart rate (QTc) ≤480 ms (Fridericia's formula).
  * Baseline oxygen saturation on room air ≥ 92%
  * Albumin ≥ 3.0 g/dL
* Women of child-bearing potential (WOCBP), defined as a sexually mature woman who has not undergone surgical sterilization or who has not been naturally postmenopausal for at least 12 consecutive months must agree to use a highly effective contraceptive method
* Patients must be willing and able to sign the informed consent form, and to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Prior treatment with an ADC with a topoisomerase I (TOP1) payload.
* Active or progressing brain metastases or evidence of leptomeningeal disease. Stable/treated brain metastases are permitted (defined as history of brain metastases previously treated with surgical resection or stereotactic radiosurgery, stable on baseline screening study MRI brain for at least 2 months (compared to comparator MRI brain) and asymptomatic without requirement for steroids or antiseizure medications.
* Persistent toxicities from previous systemic antineoplastic treatments of Grade >1, excluding alopecia and vitiligo.
* Systemic antineoplastic therapy or prohibited co-medications within 5 half-lives or 4 weeks, whichever is shorter, prior to first dose of the study drug, including investigational agents.
* Wide-field radiotherapy (e.g., >30% of marrow-bearing bones) within 4 weeks, or focal radiation with palliative intent outside the field of measurable disease within 2 weeks prior to first dose of the study drug.
* Major surgery within 4 weeks prior to first dose of study drug, or no recovery from side effects of such intervention.
* Has had clinically significant lung disease requiring systemic corticosteroid treatment within the last 6 months of randomization/registration (e.g., interstitial pneumonia, pneumonitis, pulmonary fibrosis, and severe radiation pneumonitis) or who are suspected to have such diseases by imaging at screening period.
* Patients with acute or chronic pancreatitis and/or liver cirrhosis except well compensated cirrhosis (Child-Pugh class A).
* Hepatic insufficiency manifesting as clinical jaundice, hepatic encephalopathy, and/or variceal bleed within 60 days prior to study entry.
* History of liver transplant.
* Prior allogeneic bone marrow transplantation.
* Significant cardiac disease, such as recent (within 6 months prior to first dose of the study drug) myocardial infarction or acute coronary syndromes (including unstable angina pectoris), congestive heart failure (New York Heart Association class III or IV), uncontrolled hypertension, uncontrolled cardiac arrhythmias, severe aortic stenosis.
* History of thromboembolic or cerebrovascular events, including transient ischemic attacks, cerebrovascular accidents, deep vein thrombosis, or pulmonary emboli within 3 months prior to first dose of the study drug.
* Acute and/or clinically significant bacterial, fungal, or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV).

  * Note: patients with chronic HBV, HCV or HIV infection will be eligible if they are considered upon a mutual agreement of the Investigator and the Medical Monitor as safe for enrollment and meet one of the following additional conditions:
  * Patients with HIV infection are on an established antiretroviral therapy for at least 4 weeks, and have CD4+ T-cell counts ≥350 cells/µL and HIV viral load <50 copies/mL,
  * Patients with serologic evidence of chronic HBV infection receive concurrent anti-HBV therapy and have HBV viral load below the limit of quantification,
  * Patients with a history of HCV infection must have completed curative anti-HCV therapy and have HCV viral load below the limit of quantification,
  * Patients on concurrent anti-HCV therapy have HCV viral load below the limit of quantification.
* Known or suspected allergy to the study drug or any component of the study drug.
* Concurrent participation in another investigational clinical trial.
* Pregnant or breast-feeding females.
* Prior history of malignancy other than inclusion diagnosis within 3 years prior to first dose of the study drug.

  * Note: excluding patients with adequately treated basal cell or squamous cell skin cancer, non-invasive superficial bladder cancer, in situ cervical cancer, in situ breast cancer, and in situ prostate cancer. Other malignancies with low risk of recurrence may also be considered following discussion with the Medical Monitor.
* Any other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with the study participation or the study drug administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for enrollment in this study.
* Chest irradiation within 1 year prior to first dose of study drug.
* Gastrointestinal obstruction or radiographic evidence of gastrointestinal obstruction within 4 weeks prior to the first dose of study drug.
* Vaccination with a live vaccine ≤30 days prior to first dose of study drug.
* Use of a strong cytochrome P450 (CYP)3A4 or CYP1A2 inducer or inhibitor ≤14 days prior to first dose of study drug or inability to discontinue use of a strong CYP3A4 or CYP1A2 inducer or inhibitor for the duration of the study.
* Ascites requiring frequent paracentesis for symptomatic management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Characterize the safety and tolerability of CUSP06 (Phase 1a and 1b) | 36 months
  Type, incidence, and severity of adverse events (AEs) and serious adverse events (SAEs) using the NCI CTCAE v.5.0.
  Frequency and duration of dose interruptions and reductions.
Determine the recommended dose for expansion (RDE) of CUSP06 (Phase 1a) | 15 months
Evaluate preliminary efficacy of CUSP06 as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (Phase 1b) | 16 months
  ORR: proportion of patients achieving a best overall response of confirmed partial or complete response (PR+CR)

SECONDARY OUTCOMES:
Evaluate the pharmacokinetic (PK) profile of CUSP06 - maximum concentration (Cmax) (Phase 1a and 1b) | 36 months
Evaluate the pharmacokinetic (PK) profile of CUSP06 - time to Cmax (Tmax) (Phase 1a and 1b) | 36 months
Evaluate the pharmacokinetic (PK) profile of CUSP06 - area under the curve (AUC) (Phase 1a and 1b) | 36 months
Evaluate the pharmacokinetic (PK) profile of CUSP06 - terminal half-life (t1/2) (Phase 1a and 1b) | 36 months
Objective response rate (ORR) as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (Phase 1a) | 18 months
  ORR is defined as proportion of patients achieving a best overall response of confirmed partial or complete response (PR+CR)
Disease control rate (DCR) as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (Phase 1a and 1b) | 36 months
  DCR is defined as disease control rate based on best overall response.
Clinical benefit rate (CBR) as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (Phase 1a and 1b) | 36 months
  CBR is defined as proportion of subjects achieving a best overall response of confirmed partial or complete response, or durable stable disease.
Duration of response (DoR) as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (Phase 1a and 1b) | 36 months
  DoR is defined as time from the date of the first documented CR/PR until first documentation of disease progression or death, whichever comes first.
Time to progression (TTP) as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (Phase 1a and 1b) | 36 months
Progression free survival (PFS) as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (Phase 1a and 1b) | 36 months
  PFS is defined as time from the date of the first dose to the date of the first documentation of disease progression or death, whichever comes first.
Overall survival (OS) as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (Phase 1a and 1b) | 42 months
  OS is defined time from the first dose date to the date of death from any cause.
For PROC patients: proportion of patients with a change from baseline CA-125 level ≥50% for at least 28 days (Phase 1a and 1b) | 36 months
Evaluate the immunogenicity of CUSP06 (Phase 1a and 1b) | 36 months
  Assessment of antidrug antibodies (ADAs)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (14):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - START Midwest, Grand Rapids, Michigan
  - NYU Cancer Institute Clinical Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - SCRI Oncology Partners, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, Houston, Texas
  - START San Antonio, San Antonio, Texas
  - NEXT Oncology, Fairfax, Virginia
- Mater Cancer Care Centre, South Brisbane, Queensland, Australia